CLINICAL TRIAL: NCT01885572
Title: National, Multicenter Post-market Surveillance Study "Patient Reported Outcome" in Breast Reconstruction Following Mastectomy With Titaniferously Coated Polypropylene Mesh (TiLOOP Bra)
Brief Title: National, Multicenter PMS Study "Patient Reported Outcome" in Breast Reconstruction Following Mastectomy With TiLOOP Bra
Acronym: PRO-BRA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pfm Medical Mepro Gmbh (Industry)
Collaborators: pfm medical gmbh (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: pfm 12k001 TiLOOP Bra
Record Dates: First submitted 2013-05-24; First posted 2013-06-25 (Estimated); Last update posted 2021-09-20 (Actual); Status verified 2021-09

CONDITIONS: Breast Reconstruction After Mastectomy
Keywords: breast reconstruction; mastectomy; mesh; breast cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TiLOOP Bra (Other): Treatment with TiLOOP Bra
  Interventions: Device: TiLOOP Bra

INTERVENTIONS:
Device: TiLOOP Bra — Titaniferously coated polypropylene mesh

SUMMARY:
This multicentre, non-randomised, observational clinical device investigation will be performed to obtain postmarketing information on the TiLOOP® Bra and in particular on the improvement of the patients' quality of life as well as on the rate of complications of the device under investigation.

The objective of this clinical investigation is to establish the feasibility, efficacy and safety of the TiLOOP® Bra.

ELIGIBILITY:
Inclusion Criteria:

The TiLOOP®Bra is designed to assist oncologically indexed skin sparing mastectomy or subcutaneous mastectomy with preservation of the nipple-areola-complex during primary breast reconstruction, secondary breast reconstruction or corrective breast surgery. Patients shall be included if they meet all of the following criteria:

Clinical Criteria (reason):

* women with indication of prophylactic operation or oncoplastic operation with support of a mesh implant
* women with histologically confirmed breast cancer or precancerosis or genetic pre-existing conditions with increased risk of breast cancer or with a family history
* the health of women must comply with ECOG (Eastern Cooperative Oncology Group) performance status 0-2

Study-related inclusion criteria - Legal reasons:

* Patient is mentally able to understand the nature, aims, or possible consequences of the clinical investigation
* Patient information has been handed out and all written consents are at hand.
* Patient is between 18 and 70 years old.

Exclusion Criteria:

Patients must be excluded if any of the following conditions exist or cannot be excluded:

Device-related exclusion criteria (contraindications):

Pathological or physical condition precluding such as:

* Pregnancy or breast-feeding patients
* Known intolerance to the mesh-implants under investigation.

Study-related exclusion criteria - Medical reasons:

* metastatic breast cancer
* medicamentous regulated diabetes with blood sugar level >250
* inadequate bone marrow function with neutrophil granulocytes <1500 and blood plates < 10000/µl
* patient with known contraindication to mesh-implants or plastic-reconstructive breast operations

Study-related exclusion criteria - Legal reasons:

* Lack of written patients informed consent.
* Lack of patient compliance regarding data collection, treatment or follow-up investigations in the scope of the protocol.
* Patient is institutionalized by court or official order (MPG§20.3).
* Participation in another operative clinical investigation.

It is thought that the study-related exclusion criteria will not significantly influence the sample of the population under investigation.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 267 (Actual)
Dates: Start 2013-11 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2021-06 (Actual)

PRIMARY OUTCOMES:
PRO | 12 months after breast reconstruction
  Measurement of the Patient Reported Outcome (PRO).

SECONDARY OUTCOMES:
PRO | 6 and 24 months after breast reconstruction
  Measurement of the Patient Reported Outcome
Complication Rate | after 6, 12 and 24 months
  Complication rate of the first 60 patients in the 6 month follow-up and of all patients after 6, 12 and 24 months.
Cosmetic Success | 6, 12 and 24 months after breast reconstruction
  Cosmetic success confirming the reinforcement will be assessed by the patient and an independent professional at a photo. The questions posed are part of the validated Breast Q questionnaire.
PRO and Complication Rate | 48 months after breast reconstruction
  Measurement of the Patient Reported Outcome and complication rate of all patients

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Paepke, MD, Principal Investigator — Technical University Munich, Ismaningerstrasse 22, 81675 Munich, Germany
Locations (8):
- Germany (8):
  - Charite Campus Mitte and Benjamin Franklin, Berlin
  - St. Gertrauden Krankenhaus, Berlin
  - Vivantes Kliniken am Urban, Berlin
  - Helios Kliniken, Berlin
  - St. Elisabeth Krankenhaus, Cologne
  - Agaplesion Markus Krankenhaus, Frankfurt am Main
  - Universitätsklinikum Schleswig-Holstein, Klinik für Frauenheilkunde, Lübeck
  - Technische Universität, München

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Thill M, Faridi A, Meire A, Gerber-Schafer C, Baumann K, Blohmer JU, Mau C, Tofall S, Nolte E, Strittmatter HJ, Ohlinger R, Paepke S. Patient reported outcome and cosmetic evaluation following implant-based breast-reconstruction with a titanized polypropylene mesh (TiLOOP(R) Bra): A prospective clinical study in 269 patients. Eur J Surg Oncol. 2020 Aug;46(8):1484-1490. doi: 10.1016/j.ejso.2020.04.009. Epub 2020 Apr 15. PMID 32336622
- [Result] Nolte E, Klein E, Paepke S. Pregnancy following Unilateral Immediate Breast Reconstruction with Titanized Polypropylene Mesh (TiLOOP(R) Bra) without Compromising the Result. Plast Reconstr Surg Glob Open. 2018 Sep 14;6(9):e1919. doi: 10.1097/GOX.0000000000001919. eCollection 2018 Sep. PMID 30349788